CLINICAL TRIAL: NCT04025060
Title: Investigating Withdrawal Symptoms as Barriers to Reducing Sugar-sweetened Beverage Consumption Among Children
Brief Title: Reducing Sugar-sweetened Beverage Consumption Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NCR191271
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Pediatric Obesity; Diet, Food, and Nutrition
Keywords: sugar-sweetened beverages; caffeine withdrawal; beverages; obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Carbonated Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine-free Soda (Experimental): Consumption of caffeine-free soda daily for two weeks
  Interventions: Behavioral: Commercially-available caffeine-free soda
- Carbonated Water (Experimental): Consumption of unsweetened, carbonated water daily for two weeks
  Interventions: Behavioral: Carbonated water
- Regular Soda (Active Comparator): Consumption of regular soda daily for two weeks
  Interventions: Behavioral: Regular soda

INTERVENTIONS:
Behavioral: Commercially-available caffeine-free soda — Subjects are asked to consume caffeine-free soda daily for two weeks
  Arms: Caffeine-free Soda
Behavioral: Carbonated water — Subjects are asked to consume unsweetened, carbonated water daily for two weeks
  Arms: Carbonated Water
Behavioral: Regular soda — Subjects are asked to consume regular soda daily for two weeks
  Arms: Regular Soda

SUMMARY:
Lowering sugar-sweetened beverage (SSB) consumption is a central component of lifestyle behavior change aimed at preventing and managing obesity, yet effective reduction of SSB intakes has been met with many challenges. While their palatability, accessibility, publicity, affordability, and social acceptability contribute to frequent and sustained SSB consumption, their caffeine and sugar content may further encourage continued intake. Although adverse health consequences of excessive SSB consumption are well documented, the extent to which their pleasant taste (due primarily to their sugar content) and post-ingestive effects (due to their sugar and/or caffeine content) positively reinforce consumption among children has not been elucidated. The purpose of this study is to conduct a pilot intervention to examine the feasibility of removing caffeinated SSBs from the child diet and to explore whether caffeinated SSB removal induces withdrawal symptoms in 8-11 (3rd-5th grade) year old children. Participants will be randomly assigned to replace their usual caffeinated SSB consumption with either caffeinated SSBs, caffeine-free SSBs or sparkling water provided by the study team for two weeks.

DETAILED DESCRIPTION:
Sugar-sweetened beverages (SSBs) significantly contribute to sugar and calorie intakes, and their consumption is associated with metabolic disease. Sweetened beverages also account for the majority of pediatric caffeine consumption. It is well-established that habitual caffeine use leads to dependence in adults and evidence for sugar dependence has been documented. However, caffeine and/or sugar dependence related to sweetened beverage consumption has not been evaluated, and determinants of their consumption among youth are severely understudied. It is critical to elucidate whether they may be physiologically or psychologically dependent on these beverages, particularly SSBs, which contain both caffeine and sugar.

The purpose of this study is to conduct a pilot study where caffeinated SSB's are replaced with caffeinated SSBs provided by the study team (control) or with caffeine-free and unsweetened alternatives (also provided by the study team) for 2 weeks, among children who habitually consume caffeinated SSBs.

Lowering SSB consumption is a central component of lifestyle behavior change aimed at preventing and managing obesity, yet effective reduction of SSB intakes has been met with many challenges. While their palatability, accessibility, publicity, affordability, and social acceptability contribute to frequent and sustained SSB consumption, their caffeine and sugar content may further encourage continued intake. Although adverse health consequences of excessive SSB consumption are well documented, the extent to which their pleasant taste (due primarily to their sugar content) and post-ingestive effects (due to their sugar and/or caffeine content) positively reinforce consumption among children has not been elucidated. This is particularly important to study among children from low-income and minority backgrounds, as these children have the highest rates of SSB intake and the highest prevalence of obesity.

Specific Aims and Hypotheses:

1. Examine the feasibility of an intervention to remove caffeinated SSB from the child diet. We hypothesize that caffeinated SSB avoidance will be feasible among children, but that compliance will be lowest among those assigned to sparkling water, devoid of both caffeine and sugar. Compliance with beverage assignments will be assessed using daily online questionnaires and weekly dietary recalls.
2. Explore the extent to which caffeinated SSB removal induces withdrawal symptoms. We hypothesize that replacement of caffeinated SSBs with caffeine-free SSBs, or sparkling water will induce withdrawal symptoms compared to control (usual caffeinated SSB consumption). Participants will complete a child-adapted version of the validated Caffeine Withdrawal Symptoms Questionnaire (CWSQ) at baseline and daily (online) during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Reports regular consumption of caffeinated sugar-sweetened beverages, defined as consuming ≥ 12 ounces of caffeinated SSB's per day

Exclusion Criteria:

* Poorly managed chronic medical condition; current or prior eating order diagnosis; asthma requiring medication in past three months; history of migraines; regular consumption (≥ 1 serving per week) of other caffeinated beverages, such as energy drinks, regular coffee, or hot tea

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Adherence | Two weeks
  Adherence will be assessed by summing the number of study beverages consumed each day over the course of the intervention.
Withdrawal Symptoms | Average withdrawal scores over first 72 hours of intervention
  We will assess caffeine withdrawal symptoms using a child-adapted version of the validated caffeine withdrawal symptoms questionnaire (CWSQ). Participant responses to the CWSQ are on a Likert scale, where a score of "0" is not at all and "4" is "extremely"

CONTACTS AND LOCATIONS:
Locations (1):
- Milken Institute School of Public Health and GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04025060/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04025060/SAP_001.pdf